CLINICAL TRIAL: NCT04215796
Title: Evaluation of the Safety, Usability and Efficacy of the ReX-C® System in Medication Management, in Patients Receiving CFTR Modulators (Kalydeco, Orkambi and/or Symdeko) for the Treatment of Cystic Fibrosis (CF).
Brief Title: Evaluation of the ReX-C System, in Patients Receiving CFTR Modulators for the Treatment of Cystic Fibrosis (CF).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dosentrx Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXC-054-2019-CLE
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Cystic Fibrosis; Adherence, Medication
MeSH Terms: conditions — Cystic Fibrosis; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Open study for subjects receiving home-based medication: CFTR modulators (Kalydeco, Orkambi, Simdeko) treatment. Subjects receive these medication by ReX-C device. Medication adherence, treatment instructions and side effects are recorded and monitored online in real time during the Study, by the ReX-C system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReX-C intervention (Experimental): Subjects use ReX-C to receive CFTR modulators medications. Adherence data, side effects and response to treatment are monitored online in real time via ReX-C cloud.
  Interventions: Device: ReX-C system

INTERVENTIONS:
Device: ReX-C system — CFTR modulators are dispensed to patients via ReX-C system

SUMMARY:
Cystic fibrosis (CF) is a progressive multisystem disorder characterized by abnormalities in the transport of chloride ions in human airway epithelial cells, leading to frequent lung infections, decreased pulmonary function, inability to properly digest food and absorb essential nutrients, and complications with many organs.

Patients with CF spend hours daily, in treatments required to manage their disease, including hours of physiotherapy and inhalation and treatment with many daily pills. CF treatment load heavy burden on patients and families and the inevitable consequence of these treatment demands is widespread non-adherence to therapy.

CFTR modulators (trade name Kalydeco, Orkambi, Simdeco) is a highly efficient drug approved to treat CF in patients with certain mutations. It is the first drug that treats the underlying cause rather than the symptoms of the disease. It is also one of the most expensive drugs, costing over $300,000 per patient per year. Despite of its proven efficacy and approved reimbursement for certain patients, non-adherence is common among CF patients, resulting from the heavy burden of daily treatment required to manage CF disease.

DETAILED DESCRIPTION:
ReX is a hand-held, mobile device intended to provide solid oral medication on patient's demand according to a pre-programmed treatment protocol. ReX addresses poor patient adherence, tracks patient's response to treatment and enhances patient engagement to therapy. The system comprises a reusable drug dispensing unit (Dispenser), a disposable Cassette containing the prescribed medication, a cellphone app, and the ReX cloud. The Dispenser manages pill administration. It includes a touch screen which guides the user and presents patient-specific clinical surveys and therapy information. The Dispenser contains a chargeable battery and indicators demonstrating device and battery status; a pill window enabling pills to be viewed; operational sensors; and communication to an app on cellphones. The patient receives the Cassette from the pharmacy, pre-filled with his/her specific medication. The Cassette is inserted into the Dispenser where it is locked in place. All therapy and patient survey data are transferred to a patient-specific domain on DosentRx' proprietary web-based cloud, named ReX cloud.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, at least 12 years of age
2. Subject is able to swallow pills and during training successfully achieves 2 administrations of "demo" pills (Tic-Tac sweets) by ReX-C.
3. Subject is able to read and understand the Informed Consent Form.
4. Subject was diagnosed with CF and receives CFTR modulators medication.
5. Subject is intended to receive Kalydeco OR Orkambi OR Symdeko during the 12 months study period.
6. Subject takes medication therapy at home.
7. Subject is fluent in one of the following languages: Hebrew, Arabic.

Exclusion Criteria:

1. Subject has significant physical disability including; poor fine motor skills, impaired visual or auditory faculties, mental disorders or other impairment affecting ability to provide Informed Consent or use the ReX-C dispensing unit effectively.
2. Subject failed to extract 2 "demo" pills during ReX-C training.
3. Subject is participating in another clinical study that does not permit participation in two studies simultaneously.
4. Subject is at end stage or terminal illness with anticipated life expectancy of 6 months or less.

   -

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of safety events during administration of oral oncolytic medications by ReX-C | 12 months
  Safety events include: pill overdose, pill inhalation during pill ingestion, pill malformation upon dispensing and any severe adverse events related to pill intake by the ReX-C device.
Rate of subjects feel comfortable to use ReX-C for pill intake and medication managment and define the system as "Easy to use" | 12 months
  At least 70% of subjects:
  A. Complete at least 6 months with Rex-C. B. Define the system as easy to use and are willing to continue using it for their medication treatment.
Rate of adherence (number of pill intakes) during treatment with ReX-C | 12 months
  A. Adherence rate when using the ReX-C system is > 80%.
  B. Adherence rate is enhanced by the following measures:
  * At least 80% of missed/ delayed doses recorded by ReX-C are subsequently taken by subjects following real-time reminder communication.
  * Subject's self-report by adherence questionnaire

SECONDARY OUTCOMES:
Rate of improvement in patients health condition when using ReX-C compared with historical data of the same subject, taking identical CFTR modulator in the conventional way | 24 months (12 months historical data, before study initiation), 12 months ReX intervention
  Improvement of 10-20% in the following parameters, compared between period of ReX intervention versus historical period when same medication was taken in the conventional way.
  A. Reduced # of acute exacerbation B. Improved PFT C. Reduced hospitalization events D. Decreased antibiotic treatment events

CONTACTS AND LOCATIONS:
Overall Officials: David Shoseyyov, MD, Principal Investigator — Hadassah Medical Center, Pediatric department, Jerusalem, Israel; Galit Livnat-Levanon, MD, Principal Investigator — Pediatric unit, Lady Davis Carmel Medical Center, Haifa, Israel
Locations (2):
- Israel (2):
  - Hadassah Medical Organization, Jerusalem, Select One
  - Carmel Medical Center, Haifa